CLINICAL TRIAL: NCT06439368
Title: Effect of Dezocine Combined With Sufentanil on the Quality of Postoperative Recovery and Analgesic Effect in Patients Undergoing Thoracic Surgery: a Randomized, Double-blind, Parallel-controlled, Multicenter Clinical Study
Brief Title: Effect of Dezocine Combined With Sufentanil on the Quality of Postoperative Recovery and Analgesic Effect in Patients Undergoing Thoracic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yangtze River Pharmaceutical Group Co., Ltd. (Industry)
Collaborators: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NFEC-2023-005
Record Dates: First submitted 2024-05-08; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Rehabilitation; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — dezocine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): At the end of the operation, dezocine 1.0 mg/kg + sufentanil 2.0 ug/kg (prepared as 200 ml, background volume 2 ml/h, single dose 2 ml/time, locking time 15 min) was uniformly administered by PCIA; 3 ml test dose was administered immediately after the analgesic pump was connected at the end of the operation, and continuous analgesia was performed for 48 hours after the operation.
  Interventions: Drug: Dezocine
- Control group (Other): At the end of the operation, sufentanil injection 3.0 ug/kg (prepared as 200 ml, background volume 2 ml/h, single dose 2 ml/time, locking time 15 min) was uniformly administered by PCIA; 3 ml test dose was immediately administered after the analgesic pump was connected at the end of the operation, and continuous analgesia was performed for 48 hours after the operation.
  Interventions: Drug: Dezocine

INTERVENTIONS:
Drug: Dezocine — At the end of the operation, dezocine 1.0 mg/kg + sufentanil 2.0 ug/kg (prepared as 200 ml, background volume 2 ml/h, single dose 2 ml/time, locking time 15 min) was uniformly administered by PCIA; 3 ml test dose was administered immediately after the analgesic pump was connected at the end of the operation, and continuous analgesia was performed for 48 hours after the operation.
  Other Names: sufentanil

SUMMARY:
The goal of this clinical trial is to evaluate the effect of dezocine combined with sufentanil on postoperative recovery quality and analgesic effect in patients undergoing thoracic surgery. It will also learn about the safety of dezocine. Researchers will compare drug dezocine to Sufentanil to see if dezocine works to Improve postoperative pain and recovery quality for patients. Participants will undergo elective surgery and receive PCIA postoperatively，taking dezocine combine with sufentanil,or only sufentanil respectively. Visit the VAS score after connecting the analgesic pump 24h and 48h，and evaluate the Quality of Recovery

-15 score.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective thoracoscopic surgery under general anesthesia, and patients with moderate to severe pain requiring opioids or opioid-non-opioids combined analgesia after surgery as assessed by the investigator;
2. 18 to 65 years of age, male or female;
3. Body mass index (BMI) between 18-30 kg/m ² (BMI = body weight (kg)/height ² (m ²)), including borderline values;
4. Modified Mahalanobis score < III;
5. ASA grade I ~ III;
6. Voluntarily signed informed consent.

Exclusion Criteria:

1. Inability to understand the nature, significance, possible benefits, possible inconveniences and potential risks of the trial, or inability to understand the study procedures and pain-related assessment methods;
2. Patients who cannot accept the postoperative analgesia specified in the protocol;
3. Clinician judgment: liver and kidney dysfunction has clinical significance (ALT and AST > 2 times the upper limit of normal; BUN and/or Urea > 2 times the upper limit of normal, Cr > 2 times the upper limit of normal; dialysis treatment within 28 days before surgery), or coagulation dysfunction has clinical significance (PT or APTT or TT > the upper limit of normal), or poor blood pressure control (sitting SBP > 160 mmHg or SBP < 90 mmHg), or oxygen saturation (without oxygen) < 94%;
4. Patients with high risk of respiratory depression or respiratory depression (such as sleep apnea syndrome);
5. Patients who are allergic to the test drugs (dezocine, sufentanil);
6. History of bronchial asthma;
7. Patients with hypothyroidism;
8. Patients with uncontrolled gastrointestinal ulcers, gastrointestinal bleeding or perforation before surgery; or patients with paralytic ileus;
9. Patients with chronic (continuous 3 months or intermittent up to 6 months) pain associated with non-surgical sites;
10. Craniocerebral injury, possible intracranial hypertension, cerebral aneurysm, cerebrovascular accident history or suffering from central nervous system diseases (such as epilepsy);
11. Suffering from mental system diseases (such as depression), or long-term use of psychotropic drugs;
12. Patients who cannot evaluate the pain intensity after surgery or are transferred to ICU;
13. Evidence of severe cardiac dysfunction (NYHA class III and IV), unstable angina pectoris or acute myocardial infarction within 6 months before enrollment;
14. Estimated operative blood loss greater than 1000 ml or other serious complications during surgery;
15. Patients with a history of drug abuse, drug abuse and alcohol abuse within 2 years before the start of the screening period; Alcohol abuse was defined as regular consumption of more than 14 drinks/week (1 drink = 150 mL wine or 360 mL beer or 45 mL spirits);
16. Patients who have been taking opioids for a long time (continuous use for 1 month or intermittent use for up to 3 months), or who are tolerant to opioids;
17. Patients who have used monoamine oxidase inhibitors within 2 weeks;
18. Participating in any clinical trial as a subject within 3 months;
19. Pregnant or lactating women or patients with fertility plan within 6 months (including men);
20. Patients who are judged unsuitable for participation by other investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
QoR-15 score at 24 hours after connection to analgesic pump | 24 hours
  QoR-15 is Quality of recovery-15,score ranges from 0 (QoR extremely poor) to 150 (QoR extremely good)

SECONDARY OUTCOMES:
QoR-15 score at 48 hours after connection to analgesic pump | 48 hours
  QoR-15 is Quality of recovery-15,score ranges from 0 (QoR extremely poor) to 150 (QoR extremely good)
Proportion of patients with ≥ 8 points increase in QoR-15 score from baseline at 24hours and 48hours after connection to analgesic pump | 24 hours and 48 hours
  QoR-15 is Quality of recovery-15,score ranges from 0 (QoR extremely poor) to 150 (QoR extremely good)
Patient global impression of change score at 48 hours after connection to analgesia pump | 48 hours
Static NRS score at 2hours, 4hours, 6hours, 12hours, 24hours, 36hours, 48hours after connection to analgesia pump | 2hours, 4hours, 6hours, 12hours, 24hours, 36hours, 48hours
Number of effective compressions of analgesic pump with in 48 hours after connection of analgesic pump | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kexuan Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Yes